CLINICAL TRIAL: NCT06599411
Title: Identification Des Marqueurs Biologiques cutanés et Sanguins prédictifs de réponse Aux Traitements systémiques au Cours Des Maladies cutanées Inflammatoires Chroniques
Brief Title: Identification of Cutaneous and Blood Biomarkers Predictive of Response to Systemic Treatments During Chronic Inflammatory Skin Diseases
Acronym: ImmuneSkinBank
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240183
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Atopic Dermatitis; Psoriasis; Hidradenitis Suppurativa; Lichen Planus; Cutaneous Lupus; Dermatomyositis; Cutaneaous Scleroderma; Neutrophilic Dermatosis; Cutaneous Granulomatosis; Active Leprosy
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis; Hidradenitis Suppurativa; Lichen Planus; Dermatomyositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Affected by inflammatory skin disease
  Interventions: Other: Sampling
- Controls: Plastic surgery patients who have had any type of surgery resulting in healthy skin remnants
  Interventions: Other: Sampling

INTERVENTIONS:
Other: Sampling — Collection of an additional volume of blood Superficial skin biopsy Skin swab
  Groups: Patients
Other: Sampling — Collection of an additional volume of blood Preservation of post-operative skin remnants Skin swab
  Groups: Controls

SUMMARY:
Chronic inflammatory skin diseases constitute a heterogeneous group of pathologies. They affect the skin but also other organs (joints, lungs, muscles, etc.). Their prognosis and response to treatments is extremely variable. The discovery of prognosis factors will help to precisely guide the treatment regimen and its intensification based on individual markers. The identification of new therapeutic targets is essential to develop new innovative treatments for inflammatory skin diseases.

The main objective is to identify new cellular or molecular prognostic factors associated with treatment response at 1 year in inflammatory skin diseases.

The secondary objectives are a better understanding of the pathophysiology of chronic inflammatory skin diseases, the identification of new cellular, molecular and microbiological prognostic factors associated with the clinical state after 10 years of evolution and the identification of prognostic markers of drug toxicity.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Age>18 years
* Informed consent signed by the patient
* Diagnosis of moderate to severe chronic inflammatory skin disease (IGA score 3 or 4) including: atopic dermatitis, psoriasis, hidradenitis suppurativa, lichen planus, cutaneous lupus, dermatomyositis, cutaneous scleroderma (=morphea), neutrophilic dermatosis, cutaneous granulomatosis
* Or diagnosis of active leprosy (tuberculoid, lepromatous, reversion type 1, reversion type 2, hypersensitivity type 3), excluding pure neurological leprosy. Classification into 5 stages according to the Ridley and Jopling classification [1], Reversion reaction (type 1 reaction) and leprous erythema nodosum (type 2 reaction).

Healthy controls :

* Age>18 years
* Plastic surgery patients who have had any type of surgery resulting in healthy skin remnants
* Informed consent signed by the patient
* Absence of known cutaneous or systemic inflammatory disease.

Exclusion Criteria:

* Under guardianship or curatorship
* Pregnant or breastfeeding woman
* Lack of affiliation with a social security system
* Systemic treatment in progress or received less than 3 months ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients affected by inflammatory skin disease and controls
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2035-10-01 (Estimated); Study Completion 2044-10-01 (Estimated)

PRIMARY OUTCOMES:
Therapeutic response | At 1 year
  It is defined as complete or partial remission on the Investigator/Physician Global Assessment (IGA/PGA) scale.

SECONDARY OUTCOMES:
Expression of markers of blood and skin immunological signaling pathways | At inclusion
  Mainly Th1, Th2, Th9, Th17, Th22 and Treg
Expression of markers of blood and skin immunological signaling pathways | At 4 months
  Mainly Th1, Th2, Th9, Th17, Th22 and Treg
Expression of markers of blood and skin immunological signaling pathways | At 1 year
  Mainly Th1, Th2, Th9, Th17, Th22 and Treg
Expression of markers of blood T cell populations and skin transcriptomics | At inclusion
Expression of markers of blood T cell populations and skin transcriptomics | At 4 months
Expression of markers of blood T cell populations and skin transcriptomics | At 1 year
Therapeutic response | At inclusion
  Based on markers of blood T cell populations and skin transcriptomics
Therapeutic response | At 4 months
  Based on markers of blood T cell populations and skin transcriptomics
Therapeutic response | At 1 year
  Based on markers of blood T cell populations and skin transcriptomics
Therapeutic response | At 2 years
  Based on markers of blood T cell populations and skin transcriptomics
Therapeutic response | At 3 years
  Based on markers of blood T cell populations and skin transcriptomics
Therapeutic response | At 4 years
  Based on markers of blood T cell populations and skin transcriptomics
Therapeutic response | At 5 years
  Based on markers of blood T cell populations and skin transcriptomics
Therapeutic response | At 6 years
  Based on markers of blood T cell populations and skin transcriptomics
Therapeutic response | At 7 years
  Based on markers of blood T cell populations and skin transcriptomics
Therapeutic response | At 8 years
  Based on markers of blood T cell populations and skin transcriptomics
Therapeutic response | At 9 years
  Based on markers of blood T cell populations and skin transcriptomics
Therapeutic response | At 10 years
  Based on markers of blood T cell populations and skin transcriptomics
Microbiota markers | At inclusion
  Identification of cluster specific to the pathology, identification of an over-representation of one or more microbiological species.
  For patients and controls
Microbiota markers | At 1 year
  Identification of cluster specific to the pathology, identification of an over-representation of one or more microbiological species.
  For patients only
Proportion of patients suffering from adverse effects of systemic treatments | At inclusion
  According to the CTCAE classification and MedDRA
Proportion of patients suffering from adverse effects of systemic treatments | At 4 months
  According to the CTCAE classification and MedDRA
Proportion of patients suffering from adverse effects of systemic treatments | At 1 year
  According to the CTCAE classification and MedDRA
Proportion of patients suffering from adverse effects of systemic treatments | At 2 years
  According to the CTCAE classification and MedDRA
Proportion of patients suffering from adverse effects of systemic treatments | At 3 years
  According to the CTCAE classification and MedDRA
Proportion of patients suffering from adverse effects of systemic treatments | At 4 years
  According to the CTCAE classification and MedDRA
Proportion of patients suffering from adverse effects of systemic treatments | At 5 years
  According to the CTCAE classification and MedDRA
Proportion of patients suffering from adverse effects of systemic treatments | At 6 years
  According to the CTCAE classification and MedDRA
Proportion of patients suffering from adverse effects of systemic treatments | At 7 years
  According to the CTCAE classification and MedDRA
Proportion of patients suffering from adverse effects of systemic treatments | At 8 years
  According to the CTCAE classification and MedDRA
Proportion of patients suffering from adverse effects of systemic treatments | At 9 years
  According to the CTCAE classification and MedDRA
Proportion of patients suffering from adverse effects of systemic treatments | At 10 years
  According to the CTCAE classification and MedDRA

IPD SHARING:
Plan to Share IPD: Undecided